CLINICAL TRIAL: NCT06051552
Title: Development and Validation for Muti-stage Prognostic Prediction Model in Patients With Moyamoya Disease Undergoing Revascularization Surgery
Brief Title: Prognostic Prediction Model in Patients With Moyamoya Disease Undergoing Revascularization Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor & Director, Beijing Tiantan Hospital
Other Study IDs: WXY20230918
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Moyamoya Disease
Keywords: Perioperative management; Moyamoya Disease; Predictive Model; Revascularization Surgery; Anesthesia
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Moyamoya Disease (MMD) is a rare chronic cerebrovascular disease characterized by progressive occlusion of the internal carotid artery or its major branches, with blood flow compensated by the formation of an abnormal vascular network (smoky). According to the latest national epidemiological survey in 2022, the cumulative number of new cases in the population was 47,443 in two years, with the annual incidence rate increasing year by year. The first symptoms are mainly cerebral infarction, transient ischemic attack, intracranial hemorrhage, and epileptic seizure, and the onset of the disease is concentrated in the age group of 45-54 years old, which is one of the most important causes of new strokes in middle-aged and young people and imposes a heavy medical burden on the society and the family. As one of the major causes of new strokes in young and middle-aged people, it brings a heavy medical burden to society and families. Hemodialysis has been confirmed as a standard treatment for patients with smokers' disease in large sample studies to prevent bleeding and recurrence of hemorrhage; however, there is no better consensus on which anesthetic technique to use for hemodialysis in patients with MMD. Currently, the more perfect prediction model is the postoperative collateral compensation formation prediction model for direct and indirect hemodialysis, which has the advantage of making full use of the patients' preoperative baseline variables and imaging characteristics, but the relatively insufficient inclusion of the sample size and the lack of intraoperative (vital signs, respiratory parameters, local cerebral oxygenation, etc.) and postoperative (postoperative neurological injury markers, etc.) variables included in the model limits the clinical scenarios. The lack of intraoperative (vital signs, respiratory parameters, local cerebral oxygen saturation) and postoperative (postoperative neurologic injury markers) variables limits the clinical application scenarios and is unable to guide the clinical decision-making and prognosis in the important stages of the perioperative period. This study aims to establish a prospective cohort database for MMD hemodialysis that includes perioperative anesthesia management, intraoperative treatment data, and postoperative treatment variables; to integrate preoperative, intraoperative, postoperative, and near- and long-term prognostic data from multiple sources, and to construct a perioperative multi-stage, multi-dimensional prognostic prediction model.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years.
2. Imaging-confirmed moyamoya disease (CTA, CT angiography; MRA, magnetic resonance angiography；DSA, digital subtraction angiography）for MMD patients.
3. Selective Revascularization Surgery (direct or indirect);
4. Signed informed consent by the patient or legal representative.

Exclusion Criteria:

1. patients with moyamoya syndrome due to an established secondary etiology.
2. with severe cardiopulmonary disease that, in the opinion of the investigator, makes them unsuitable for participation in this study.
3. patients with a life expectancy of less than 3 months or otherwise unable to complete this study.
4. contraindication to DSA examination, severe contrast allergy or absolute contraindication to iodine contrast;
5. women of childbearing age who have a negative pregnancy test but refuse to use effective contraception.
6. women during pregnancy or breastfeeding.
7. those who are unable to complete the study due to psychiatric disorders, cognitive or mood disorders.
8. other patients who, in the opinion of the investigator, are not suitable for enrollment in the study (indicate reason).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with moyamoya disease undergoing revascularization surgery
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | 3 consecutive days after surgery
  Postoperative assessment using 3D-CAM or CAM-ICU was performed at a fixed time slot each day for 3 consecutive days, and postoperative visits were performed at the patient's bedside from 10:00 am to 16:00 pm.
Incidence of postoperative cerebral ischemic event | 2 weeks after surgery
  categorization of cerebral ischemic complications based on typical symptoms occurring within 2 weeks after surgery, and signs of new ischemia confirmed by postoperative radiology (e.g., computed tomography (CT), CT perfusion, or diffusion-weighted imaging)

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical University, Beijing Tiantan Hospital, Beijing, China